CLINICAL TRIAL: NCT01708057
Title: A Randomised, Double-blind Placebo- and Active-controlled, Multi-centre, 6-way Cross-over, Single-dose Phase IIa Study to Investigate the Bronchodilatory and Systemic Effects of 4 Different Doses of Inhaled AZD8683 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Single-dose Study to Investigate the Effects of 4 Different Doses of Inhaled AZD8683 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D1883C00007; EudraCT number: 2012-002900-42
Record Dates: First submitted 2012-10-01; First posted 2012-10-16 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: COPD; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- 1 (Experimental): Single dose of AZD8683 50 µg
  Interventions: Drug: AZD8683
- 2 (Experimental): Single dose of AZD8683 150 µg
  Interventions: Drug: AZD8683
- 3 (Experimental): Single dose of AZD8683 300 µg
  Interventions: Drug: AZD8683
- 4 (Experimental): Single dose of AZD8683 900 µg
  Interventions: Drug: AZD8683
- 5 (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo
- 6 (Active Comparator): Single dose of tiotropium 18 µg
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: AZD8683 — AZD8683 administered via inhalation
  Arms: 1; 2; 3; 4
Drug: Placebo — Placebo administered via inhalation
  Arms: 5
Drug: Tiotropium — Tiotropium administered via inhalation
  Arms: 6

SUMMARY:
This study in Chronic Obstructive Pulmonary Disease (COPD) patients will investigate the bronchodilatory effect of AZD8683. AZD8683 will be tested versus placebo and an active comparator.

DETAILED DESCRIPTION:
A randomised, double-blind placebo- and active-controlled, multi-centre, 6-way cross-over, single-dose phase IIa study to investigate the bronchodilatory and systemic effects of 4 different doses of inhaled AZD8683 in patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures Male or female, age ≥ 40 years at Visit 1. Women must be of non-childbearing potential or must have been stable on a highly effective contraceptive method for at least 3 months prior to Visit 1 and be willing to continue until follow-up
* Clinical diagnosis of COPD for more than 1 year at Visit 1
* FEV1 ≥ 30 to < 80% of the predicted normal value (post-bronchodilator) at Visit 2 and post-bronchodilator FEV1/FVC < 70%
* Reversible airway obstruction

Exclusion Criteria:

* Significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the result of the study, or the patient's ability to participate in the study.
* An exacerbation of COPD (defined as use of oral/parenteral glucocorticosteroids (GCS) and/or antibiotics and/or hospitalisation related to COPD) within 6 weeks of Visit 1or during the enrolment period
* Treatment with systemic GCS within 6 weeks of Visit 2 or during the enrolment period
* Respiratory tract infection of clinical relevance within 30 days of Visit 4, as judged by the Investigator
* Long-term oxygen therapy, as judged by the Investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, MD, Study Director — AstraZeneca R&DMolndal, Sweden
Locations (6):
- Poland (4):
  - Bialystok
  - Lodz
  - Proszowice
  - Wroclaw
- Sweden (2):
  - Gothenburg
  - Lund

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 subjects were enrolled. Of these, 3 subjects were randomized to receive a treatment sequence consisting of 6 different treatments in random order. The study was terminated prematurely, hence only one period out of six planned was performed.
Groups:
- AFBECD: AZD8683 50 ug followed by Placebo followed by AZD8683 150 ug followed by Spiriva® 18 ug followed by AZD8683 300 ug followed by AZD8683 900 ug
- FEADBC: Placebo followed by Spiriva® 18 ug followed by AZD8683 50 ug followed by AZD8683 900 ug followed by AZD8683 150 ug followed by AZD8683 300 ug
- DCEBFA: AZD8683 900 ug followed by AZD8683 300 ug followed by Spiriva® 18 ug followed by AZD8683 150 ug followed by Placebo followed by AZD8683 50 ug
Period: Overall Study
Arm/Group | AFBECD | FEADBC | DCEBFA
Started | 1 | 1 | 1
Completed | 0 | 0 | 0
Not Completed | 1 | 1 | 1
Not completed — Withdrawal due to study termination. | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total Baseline: All Patients population
Arm/Group | Total Baseline
Number analyzed (Participants) | 3
Age, Customized [Number; unit: participants]
  <=18 year | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex/Gender, Customized [Number; unit: participants]
  Male | 2
  Female | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 3
  other | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak FEV1 (0-24h)
Description: The maximum value over 24 hours post-dose, as change from baseline
Time Frame: The first 24 hours following dose administration
Population: As the study was terminated prematurely none of the randomised patients have been analysed.
Groups:
- AZD8683 150 ug: AZD8683 150 ug via Turbuhaler + Turbuhaler Placebo +Handihaler Placebo for Spiriva
- AZD8683 300ug: AZD8683 300 ug via Turbuhaler + Turbuhaler Placebo +Handihaler Placebo for Spiriva
- AZD8683 900ug: AZD8683 900 ug via Turbuhaler + placebo for Spiriva via HandiHaler
- Spiriva 18 ug: Turbuhaler® Placebo+Handihaler® Spiriva® 18 μg
- Placebo: Turbuhaler® Placebo+Handihaler® Placebo for Spiriva®
- AZD8683 50ug: AZD8683 50 ug via Turbuhaler + Turbuhaler Placebo +Handihaler Placebo for Spiriva
Arm/Group | AZD8683 150 ug | AZD8683 300ug | AZD8683 900ug | Spiriva 18 ug | Placebo | AZD8683 50ug
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Trough FEV1 (22-26h)
Description: The average over 22 to 26 hours, as change from baseline
Time Frame: 22 to 26 hours following dose administration
Population: As the study was terminated prematurely none of the randomized patients have been analysed.
Arm/Group | AZD8683 150 ug | AZD8683 300ug | AZD8683 900ug | Spiriva 18 ug | Placebo | AZD8683 50ug
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Average FEV1 as a Change From Baseline
Description: Average FEV1 (0-24h): The average over 0 to 24 hours
Time Frame: The first 24 hours following dose administration
Population: As the study was terminated prematurely none of the randomized patients have been analysed.
Arm/Group | AZD8683 150 ug | AZD8683 300ug | AZD8683 900ug | Spiriva 18 ug | Placebo | AZD8683 50ug
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum Increase in Systolic Blood Pressure [SBP]
Description: Maximum (post-dose values - baseline value) for each treatment visit.
Time Frame: baseline, 24hr post dose
Population: As the study was terminated prematurely none of the randomised patients have bean analysed.
Arm/Group | AZD8683 150 ug | AZD8683 300ug | AZD8683 900ug | Spiriva 18 ug | Placebo | AZD8683 50ug
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Increase in Diastolic Blood Pressure [DBP]
Description: Maximum (post-dose values - baseline value) for each treatment visit.
Time Frame: The first 24 hours following dose administration
Population: As the study was terminated prematurely none of the randomised patients have bean analysed.
Arm/Group | AZD8683 150 ug | AZD8683 300ug | AZD8683 900ug | Spiriva 18 ug | Placebo | AZD8683 50ug
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Increase Heart Rate [HR]
Description: Maximum (post-dose values - baseline value) for each treatment visit.
Time Frame: baseline, 24hr post dose
Population: As the study was terminated prematurely none of the randomised patients have bean analysed.
Arm/Group | AZD8683 150 ug | AZD8683 300ug | AZD8683 900ug | Spiriva 18 ug | Placebo | AZD8683 50ug
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Maximum Increase in QTcF
Description: maximum (post-dose values - baseline value) for each treatment visit.
Time Frame: baseline, 24hr post dose
Population: As the study was terminated prematurely none of the randomised patients have bean analysed.
Arm/Group | AZD8683 150 ug | AZD8683 300ug | AZD8683 900ug | Spiriva 18 ug | Placebo | AZD8683 50ug
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: PK Parameters (AZD8683)
Description: Cmax, tmax, AUC
Time Frame: Pre-dose, 24hr post-dose
Population: As the study was terminated prematurely none of the randomised patients have bean analysed.
Arm/Group | AZD8683 150 ug | AZD8683 300ug | AZD8683 900ug | Spiriva 18 ug | Placebo | AZD8683 50ug
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 days
Groups:
- 50ug AZD8683: AZD8683 50 ug via Turbuhaler + Turbuhaler Placebo +Handihaler Placebo for Spiriva
- 150 ug AZD8683: AZD8683 150 ug via Turbuhaler + Turbuhaler Placebo +Handihaler Placebo for Spiriva
- 300 ug AZD8683: AZD8683 300 ug via Turbuhaler + Turbuhaler Placebo +Handihaler Placebo for Spiriva
- 900 ug AZD8683: AZD8683 900 ug via Turbuhaler + placebo for Spiriva via HandiHaler;
- 18ug Spiriva: Turbuhaler® Placebo+Handihaler® Spiriva® 18 μg
Arm/Group | 50ug AZD8683 | 150 ug AZD8683 | 300 ug AZD8683 | 900 ug AZD8683 | 18ug Spiriva | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0 | 0/1 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0 | 1/1 | 0/0 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50ug AZD8683 (N=1) | 150 ug AZD8683 (N=0) | 300 ug AZD8683 (N=0) | 900 ug AZD8683 (N=1) | 18ug Spiriva (N=0) | Placebo (N=1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days